CLINICAL TRIAL: NCT02504281
Title: Study on the Association Between Skewed X Chromosome Inactivation(SXCI) and Recurrent Miscarriage(RM) and the Possible Genetic Mechanism
Brief Title: Study on the Association Between SXCI and RM and the Possible Genetic Mechanism
Status: Completed | Type: Observational
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Other Study IDs: JIAI E2015-02
Record Dates: First submitted 2015-07-19; First posted 2015-07-21 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2020-05

CONDITIONS: Infertility Female; Recurrent Miscarriage
MeSH Terms: conditions — Infertility, Female; Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from the females
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RM: Women 18-43 years of age who are scheduled for IVF or ICSI with a history of recurrent spontaneous abortion (miscarriage occurred earlier than 22 weeks of gestation for equal or greater than 3 times) in our IVF institute.
- Control: Normal females who are visiting Shanghai JIAI genetics and IVF institute for IVF/ICSI because of only male factor.

SUMMARY:
To determine whether there is higher incidence of skewed X chromosome inactivation(SXCI) in the recurrent miscarriage(RM) population compared with normal population, and verify the existing hypothesis of the possible genetic mechanisms underlying the association between SXCI and RM.

DETAILED DESCRIPTION:
Recurrent spontaneous abortion (RSA), defined as 2 or more consecutive pregnancy losses before 20-22 weeks of gestation, is a multifactorial disorder that affects about 5% of all couples.In up to 50% of women who have experienced RSA, the cause still remains unexplained, with genetic problem proposed as a main cause. X chromosome inactivation (XCI) is a physiological phenomenon in female mammals for 'dosage compensation' of X-linked genes with males. A normal female is mosaic, with about one-half of her somatic cells expressing the paternal derived X and the remainder of her cells using maternal X. In some situations, however, the inactivation is not random, resulting in a female having most or even all her somatic cells inactivating the same X chromosome from either paternal or maternal resource, which is known as skewed X-chromosome inactivation (SXCI).Evidence of an association between skewed X chromosome inactivation (SXCI) and idiopathic recurrent spontaneous abortion (RSA) is conflicting. This is a single-center observational case-control trial to determine whether there is higher incidence of skewed X chromosome inactivation(SXCI) in the recurrent miscarriage(RM) population compared with normal population, and verify the existing hypothesis of the possible genetic mechanisms underlying the association between SXCI and RM.

ELIGIBILITY:
Inclusion Criteria:

* 1) regular menstrual cycles and normal level of E2, P, FSH, LH, T, RPL in the early follicular phase; 2) no history of gynecologic or other pelvic operations; 3) no history of hormone medicine application in the last 3 months; 4) no history of poison contact; 5) normal uterine and adnexal ultrasonography; 6) TORCH(-), chlamydia(-), mycoplasma(-), normal leucorrhoea routine, anti-phospholipid antibody (-), antinuclear antibody(-); 7) for the couple, no blood type incompatibility or ABO antibody IgG≤1：64 and normal blood chromosome analysis; 8) condoms are used for contraception.

Exclusion Criteria:

* 1) BMI<18.5 or >24.9; 2) hydrosalpinx without operation; endometriosis; polycystic ovary syndrome; adenomyosis; uterine leiomyomata(submucous myoma or non-submucous myoma which size was exceed 4cm and/or with the compressed endometrium);uterine cavity lesions(such as uterine malformation, intrauterine adhesions, the septate uterus, endometritis etc); 3) the former abortion is because of luteal phase defect without treatment; 4) FSH≥12IU/L or AMH<1.2ng/ml 5) thyroid dysfunction or increased CA125 level; 6) acute inflammation of genitourinary system or STD carriers; 7) unable to comply with the study procedures.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women visiting our centre for IVF/ICSI during 2015.01.01-2016.01.01 will enter RM group or control group according to their pregnant history or infertility factor.
  RM group: Women with a history of recurrent spontaneous abortion (miscarriage occurred earlier than 22 weeks of gestation for equal or greater than 2 times).
  Control group:Infertility women because of only male factor. Both groups meet the same elgibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
degree of X chromosome inactivation skewing | Within 3 months after blood collection
percentage of extremely skewed X chromosome inactivation(SXCI>90%) in each group | Within 3 months after blood collection

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, MD, Study Director — ShangHai Ji Ai Genetics & IVF Institute
Locations (1):
- Shanghai Jiai Genetics&IVF Institute, Shanghai, China

REFERENCES:
- [Derived] Sui Y, Fu J, Zhang S, Li L, Sun X. Investigation of the role of X chromosome inactivation and androgen receptor CAG repeat polymorphisms in patients with recurrent pregnancy loss: a prospective case-control study. BMC Pregnancy Childbirth. 2022 Nov 2;22(1):805. doi: 10.1186/s12884-022-05113-z. PMID 36324098